CLINICAL TRIAL: NCT04533191
Title: Binocular Custom Vision Utilizing The Light Adjustable Lens (LAL)
Status: Completed | Type: Observational
Sponsor: Vance Thompson Vision (Other)
Responsible Party: Sponsor
Other Study IDs: IIT-001
Record Dates: First submitted 2020-08-25; First posted 2020-08-31 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Cataract; Pseudophakia
MeSH Terms: conditions — Cataract; Pseudophakia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Subjects treated with LAL lens: Subjects that underwent standard of care cataract surgery and LAL IOL placement.
  Interventions: Procedure: LAL IOL lens

INTERVENTIONS:
Procedure: LAL IOL lens — Standard of care Cataract surgery with IOL placement

SUMMARY:
The objective of this investigator initiated study (IIT-001) is to obtain data on clinical methods which can be used during the examination of patients desiring binocular custom vision with the Light Adjustable Lens (LAL). An analysis of the collected data will be performed to determine whether these clinical assessments can be used by doctors to enhance their patient's clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Patients able to sign informed consent
2. Patients who plan to undergo bilateral implantation with the commercial LAL and receive binocular custom vision are eligible for study participation.

Exclusion Criteria:

* Inability to sign informed consent
* Any pathology for which, in the investigator's judgement, could reduce the subjects BCVA
* Unable to return for light treatments

Ages: 18 Years to 110 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A population of 25 patients who plan to undergo bilateral cataract surgery with implantation of commercially available Light Adjustable Lens (LAL) and receive binocular custom vision.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Binocular uncorrected distance, intermediate, and near visual acuity | Through Month one post-op
Binocular uncorrected depth of focus | Through Month one post-op

SECONDARY OUTCOMES:
Manifest refraction | Through Month one post-op
Monocular uncorrected distance visual acuity | Through Month one post-op
Monocular best corrected distance visual acuity | Through Month one post-op
Visual Satisfaction | Through Month one post-op
  Visual satisfaction will be obtained using a visual questionnaire
4th order total eye spherical aberration (Z12) | Through Month one post-op

CONTACTS AND LOCATIONS:
Locations (1):
- Vance Thompson Vision, Sioux Falls, South Dakota, United States

IPD SHARING:
Plan to Share IPD: No